CLINICAL TRIAL: NCT05327933
Title: Middle Meningeal Artery Embolization Minimizes Burdensome Recurrence Rates After Newly Diagnosed Chronic Subdural Hematoma Evacuation (MEMBRANE)
Brief Title: Preventing Recurrences of Chronic Subdural Hematoma in Adult Patients by Middle Meningeal Artery Embolization
Acronym: MEMBRANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unfallkrankenhaus Berlin (Other)
Responsible Party: Principal Investigator, Johannes Lemcke, Deputy Head Department of Neurosurgery, Unfallkrankenhaus Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMA_SP; DRKS00020465 (Other: German Clinical Trials Register)
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Hematoma, Subdural, Chronic
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery plus endovascular MMA embolization (Experimental)
  Interventions: Procedure: Surgery plus endovascular MMA embolization
- Surgery alone (Active Comparator)
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Procedure: Surgery plus endovascular MMA embolization — A micro catheter is inserted transfemorally into the branches of the middle meningeal artery (MMA) in a minimally invasive manner and the periphery is occluded using polyvinyl alcohol (PVA) particles to prevent future bleeding. If the desired catheter position cannot be achieved due to the anatomical conditions, a more proximal closure of the MMA using Onyx® or micro-electric coils is performed. Embolization of the MMA by PVA particles with sizes between 40-300 µm is preferred over embolization by coils and Onyx®, since the capillary network of the dura is entirely blocked when using particles. In order to identify the vessels to be closed, a digital subtraction angiography (DSA) is performed.
  Arms: Surgery plus endovascular MMA embolization
Procedure: Surgery alone — Evacuation of cSDH
  Arms: Surgery alone

SUMMARY:
Patients with a chronic subdural hematoma (cSDH), that is, a blood accumulation between two meninges developing over a long period of time, often have recurrent bleedings after an initial operation. The study aims to show that additional surgery reduces the risk of recurrent bleeding.

The additional procedure aims to block small blood vessels in the skull with tiny plastic particles. The small blood vessels are embolized using X-rays and a contrast medium and a fine tube that is inserted into the diseased vessels of the head via the groin.

Patients of full age who have undergone burr hole trepanation as a first operation, i.e. a blood drain through a hole in the cranial cavity, can participate in the study. Participating patients are randomly assigned to a control group with treatment according to clinical routine or a treatment group with an additional occlusion of the blood vessels in the skull. In addition, patients can consent to a genetic test to determine the relationship between a coagulation factor and the risk of recurrence of the hematoma. In order to record the test results, check-up examinations are carried out after one and three months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone surgery by means of one or more burr hole trepanations during the first manifestation of a cSDH (unihemispherical or bihemispherical) detected by computed tomography or magnetic resonance tomography
2. Age ≥18 years
3. Sufficient compliance and ability to consent
4. Patient's informed consent for surgical as well as endovascular interventional procedure and participation in the study

Exclusion Criteria:

1. Conservatively treated cSDH
2. Radiological evidence of an acute or subacute subdural hematoma, subarachnoid hemorrhage, intracerebral hematoma or epidural hematoma
3. Surgical technique: craniotomy, craniectomy, bilateral burr hole trepanation
4. Angiography cannot be performed within 72 hours after surgery
5. Age <18 years
6. Supervisory relationship
7. Pregnancy
8. Lack of informed consent
9. Lack of compliance
10. Homozygous factor XIII deficiency with residual activity <10%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
cSDH recurrence rates after surgery | Within three months of follow-up
  A recurrence occurs when at least one of the following criteria is met:
  * recurrent cSDH with at least the same volume (>- 10%) compared to the findings at baseline and / or
  * recurrent cSDH which requires surgery

SECONDARY OUTCOMES:
Impairment due to neurological deficits assessed by the modified Rankin Scale | Evaluated at three months after baseline
  Modified Rankin scale ranges from 0 (no symptoms) to 5 (severe disability)
Number of recurrence-associated complications | Within three months of follow-up
  Examined on a binary scale
Number of complications associated with interventional therapy | Within three months of follow-up
  Examined on a binary scale

OTHER OUTCOMES:
Relationship between factor XIII deficiency and risk of recurrence | Within three months of follow-up
  Factor XIII deficiency is defined if the factor XIII concentration at baseline and/or the factor XIII activity after cryopreservation is <70%.
Predisposition of the genetic variants F13A1 rs2815822 and F13B rs12134960 for factor XIII deficiency | Within three months of follow-up
  The existence of genetic variants F13A1 rs2815822 or F13B rs12134960 in the blood of the subjects is determined on a binary scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Unfallkrankenhaus Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoenning A, Lemcke J, Rot S, Stengel D, Hoppe B, Zappel K, Schuss P, Mutze S, Goelz L. Middle Meningeal Artery Embolization Minimizes Burdensome Recurrence Rates After Newly Diagnosed Chronic Subdural Hematoma Evacuation (MEMBRANE): study protocol for a randomized controlled trial. Trials. 2022 Aug 22;23(1):703. doi: 10.1186/s13063-022-06506-3. PMID 35996195